CLINICAL TRIAL: NCT02775916
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CDZ173 in Patients With Primary Sjögren's Syndrome
Brief Title: Safety, Pharmacokinetics, and Preliminary Efficacy Study of CDZ173 in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCDZ173X2203; 2014-004616-12 (EudraCT Number)
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-09

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — leniolisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDZ173 (Experimental): Capsule
  Interventions: Drug: CDZ173
- Placebo (Placebo Comparator): Capsule matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDZ173
  Arms: CDZ173
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary therapeutic efficacy of oral administrations of CDZ173 in patients with primary Sjögren's syndrome.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary therapeutic efficacy of oral administrations of CDZ173, a selective PI3K delta inhibitor, for 12 weeks, in patients with primary Sjögren's syndrome. Data from this study will provide the basis for further development of the compound for the treatment of primary Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Sjögren's syndrome (pSS)
* ESSDAI score ≥ 6 at screening visit

Exclusion Criteria:

* Secondary Sjögren's syndrome

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=324

RESULTS

PARTICIPANT FLOW:
Groups:
- CDZ173: Capsule BID
- Placebo: Capsule matching Placebo BID
Period: Overall Study
Arm/Group | CDZ173 | Placebo
Started | 20 | 10
Completed | 17 | 10
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Subject/Guardian Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDZ173 | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.85) | 44.7 (11.58) | 47.3 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Sjögren's Syndrome With Adverse Events and Death up to Day 85
Description: Safety and tolerability of CDZ173 in patients with primary Sjögren's syndrome up to End of Treatment Day 85
Time Frame: up to Day 85
Population: Safety Analysis Set - All randomized patients in the CDZ173 group (20 patients) and placebo group (10 patients) were included in the safety analysis set
Measure: Number; unit: count of participants
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
count of participants
  Participants with at least one AE | 20 | 8
  Participants with at least one SAE | 1 | 0
  Death | 0 | 0

2. Primary Outcome: Change From Baseline in the EULAR Sjögren's Syndrome Patient Reported Intensity (ESSPRI) After 12 Weeks of Treatment Day 85
Description: The ESSPRI is an established disease outcome measure for Sjögren's syndrome. The ESSPRI is a patient-reported, subjective symptom index for primary Sjögren's syndrome developed by the EULAR consortium. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight. Minimum score can be 0 and maximum score can be 10.
Time Frame: Baseline and 12 weeks (Day 85)
Population: PD analysis set - All randomized patients in the CDZ173 group (20 patients) and placebo group (10 patients) were included in the PD analysis set
Measure: Mean (Standard Deviation); unit: total score on scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on scale | -1.778 (2.4509) | -0.741 (1.3517)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = -0.69, 95% CI 2-sided [-3.343 to 1.937], Standard Deviation 1.332

3. Secondary Outcome: Change From Baseline in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) After 12 Weeks of Treatment Day 85
Description: The ESSDAI is an established disease outcome measure for Sjögren's syndrome. The instrument contains 12 organ-specific domains contributing to disease activity. For each domain, features of disease activity are scored in 3 or 4 levels according to their severity. These scores are then summed across the 12 domains in a weighted manner to provide the total score. A reduction from baseline (i.e., a negative change from baseline) in the ESSDAI score is indicative of improvement in a patient.). Each domain is assessed for activity level (i.e., no, low, moderate, high) and assigned a numerical score based on pre-determined weighting of each individual domain. An overall score is then calculated as the sum of all individual weighted domain scores. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity).
Time Frame: Baseline and 12 weeks (Day 85)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total score on scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on scale | -2.82 (1.165) | -3.34 (1.168)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.51, 95% CI 2-sided [-2.52 to 3.55], Standard Error of Mean 1.466

4. Secondary Outcome: Change From Baseline in the Short Form (36) Health Survey (SF-36) After 12 Weeks of Treatment Day 85
Description: The SF-36 is a 36-item, patient self-reported outcome measure (questionnaires) of patient health. The outcome of the questionnaires in eight scales results in two summary scores, physical component and mental component, both ranging from 0 - 100. An increase from baseline in either component summary score indicates reduced disease burden.
Time Frame: Baseline and 12 weeks (Day 85)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total score on a scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on a scale
  Physical Component Summary Score: number analyzed (Participants) | 12 | 9
  Physical Component Summary Score | 4.82 (2.235) | 4.42 (2.425)
  Mental Component Summary Score: number analyzed (Participants) | 12 | 9
  Mental Component Summary Score | 5.43 (3.415) | 1.10 (3.792)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.40, 95% CI 2-sided [-6.08 to 6.89], Standard Error of Mean 3.119
Statistical Analysis 2: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = 4.33, 95% CI 2-sided [-5.27 to 13.93], Standard Error of Mean 4.615

5. Secondary Outcome: Change in Baseline in Multidimensional Fatigue Inventory (MFI) After 12 Weeks of Treatment (Day 85)
Description: The Multidimensional Fatigue Inventory (MFI) is a patient self-reported outcome measure (questionnaires) to assess fatigue covering the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Each dimension has a possible range from 4-20. The reported total score has a range from 20-100.
  The reported total score has a range from 20-100, higher scores are associated with greater fatigue.
Time Frame: Baseline and 12 weeks (Day 85)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total score on scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on scale | -8.80 (5.557) | -2.25 (5.774)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = -6.55, 95% CI 2-sided [-21.76 to 8.66], Standard Error of Mean 7.270

6. Secondary Outcome: Change From Baseline in Physician Global Assessment of the Patient's Overall Disease Activity (Physician VAS) After 12 Weeks of Treatment Day 85
Description: A reduction from baseline (i.e., a negative change from baseline) in physician global VAS assessment score indicates improvement in patients. The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline and 12 weeks (Day 85)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total score on a scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on a scale | -10.06 (6.584) | 0.91 (7.699)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = -10.97, 95% CI 2-sided [-30.94 to 9.00], Standard Error of Mean 9.626

7. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Their Disease Activity (VAS) After 12 Weeks of Treatment Day 85
Description: A reduction from baseline (or, a negative change from baseline) in patient global VAS assessment score indicates improvement in patients.
  The visual analogue scale used is a 100 mm VAS ranging from "no disease" (0 mm) to "maximal disease activity" (100 mm).
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total score on a scale
Arm/Group | CDZ173 | Placebo
Number analyzed (Participants) | 20 | 10
total score on a scale | -4.83 (7.268) | 2.87 (8.412)
Statistical Analysis 1: Comparison: CDZ173 vs Placebo; Test type: Superiority; Mean Difference (Net) = -7.69, 95% CI 2-sided [-29.75 to 14.37], Standard Error of Mean 10.595

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit (Day 113)
Arm/Group | CDZ173 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/10
Other Adverse Events (participants affected / at risk) | 19/20 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDZ173 (N=20) | Placebo (N=10)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CDZ173 (N=20) | Placebo (N=10)
Dry Eye (Eye disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Flatulence (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Chest Discomfort (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Feeling Cold (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 1
Infected Bite (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0
Vaginal Infection (Infections and infestations) | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 7 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Sjogren's Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 10 | 1
Phlebitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT02775916/SAP_000.pdf
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02775916/Prot_001.pdf